CLINICAL TRIAL: NCT01194947
Title: Classification and Longitudinal Follow-up of Common Melanocytic Nevi With in Vivo Reflectance Confocal Microscopy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sheba Medical Center (Other Government)
Responsible Party: DR. ALONE SCOPE, SHEBA MEDICAL CENTER
Other Study IDs: SHEBA-10-8015-AS-CTIL
Record Dates: First submitted 2010-09-02; First posted 2010-09-03 (Estimated); Last update posted 2010-09-03 (Estimated); Status verified 2010-09

CONDITIONS: Common Melanocytic Nevi
Keywords: banal-appearing nevi; NEVUS
MeSH Terms: conditions — Nevus

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Study participants: patients 18 or older presenting to the Sheba Medical Center pigmented lesion clinic for skin cancer surveillance. Patients routinely undergo total skin examination that includes clinical and dermoscopic evaluation of skin lesions. Patients also routinely undergo annual total body digital photography that allows identification of new or changing lesions.
  Interventions: Device: RCM imaging

INTERVENTIONS:
Device: RCM imaging — RCM imaging will be performed using a commercially-available RCM (Vivascope 1500, Lucid Inc, Rochester, NY, USA) with 830-nm diode laser with emitting power less than 35 milliwatts

SUMMARY:
Our working hypothesis is that reflectance confocal microscopy (RCM) can identify distinct subsets of melanocytic nevi that retain their distinctive pattern over time.

ELIGIBILITY:
Inclusion Criteria:

* Patients visiting the Sheba Medical Center pigmented lesion clinic for skin examination
* Patients having at least three banal-appearing nevi, one on the upper back, one on the lower back and one on the lower extremity (excluding foot), which are amenable for RCM examination.

Exclusion Criteria:

* Patients who are unwilling or medically unable to lie down for 30 minutes.
* Pregnant women

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients visiting the pigmented lesion clinic for skin cancer surveillance
Sampling Method: Non-Probability Sample
Enrollment: 90 (Estimated)
Dates: Start 2010-09; Primary Completion 2013-09 (Estimated); Study Completion 2013-09 (Estimated)

PRIMARY OUTCOMES:
Inter-rater agreement on assignment of nevi to RCM patterns (baseline and follow-up images). | 3 YEARS

SECONDARY OUTCOMES:
Description of rates of retention and change in RCM pattern of nevi during follow-up | 3 YEARS

CONTACTS AND LOCATIONS:
Overall Officials: ALON SCOPE, MD, Principal Investigator — Sheba Medical Center
Locations (1):
- Sheba Medical Center, Rmat-gan, Israel